CLINICAL TRIAL: NCT04906005
Title: A Randomized, Double Blind, Placebo-Controlled, Single Ascending Dose Trial to Assess the Pharmacokinetics and Safety of Gadopiclenol in Japanese Healthy Volunteers Phase I Clinical Trial
Brief Title: Pharmacokinetics and Safety of Gadopiclenol in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GDX-44-013; jRCT2071210029 (Registry Identifier: jRCT (Japan Registry of Clinical Trials))
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — gadopiclenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: To ensure that administration of the IMP is carried out under double-blind conditions, an unblinded team (nurse, technician or physician) will be responsible for preparing and administrating the IMP(s). This person will ensure non-disclosure of information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gadopiclenol (Experimental): Dose per administration: dose/volume of gadopiclenol to be administered will be calculated based on patient's weight at the dose of 0.025; 0.05 or 0.1 mmol/kg BW (depending on each group).
  6 volunteers will receive gadopiclenol per group
  Interventions: Drug: gadopiclenol
- Placebo (Placebo Comparator): Dose per administration: similar dose (Volume/weight) as the one used for Gadopiclenol in the considered group.
  3 volunteers will receive gadopiclenol per group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: gadopiclenol — administration by intravenous (IV) bolus injection at 2 mL/s rate without dilution, followed by a saline flush of at least 5 mL at the same rate to ensure complete injection of the contrast agent.The gadopiclenol administration is performed by power injecto
  Arms: gadopiclenol
Drug: Placebo — intravenous (IV) bolus injection at 2 mL/s, followed by a saline flush of at least 5 mL to be in the same conditions as for gadopiclenol administration.The gadopiclenol administration is performed by power injector
  Arms: Placebo

SUMMARY:
This single center, single ascending dose, double blind, randomized, placebo-controlled phase I trial will include male and female Japanese healthy volunteers. Within a 4-week run-in period before inclusion in the trial, healthy volunteers will be checked for inclusion/non-inclusion criteria and will then be randomized and administered with gadopiclenol or placebo. For each healthy volunteer, there will be a confinement period of one night before the inclusion visit and 2 days post administration at the clinical unit. The healthy volunteers will return to the clinical unit for safety visit 7 days after study product administration.

In each dose group, 6 healthy volunteers (3 male and 3 female) will receive gadopiclenol and 3 healthy volunteers (2M/1F or 1M/2F) will receive placebo (physiological saline solution, 0.9% sodium chloride) in one single intravenous administration.

Dose escalation from one group to the next group will be sequential and will be allowed only if the clinical and biological safety of all healthy volunteers from the previous tested dose is acceptable. The decision will be made by a Trial Safety Review Board (TSRB), consisting in members of Guerbet team and the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* A Japanese healthy volunteer is defined as being born in Japan and having both parents and four grandparents (maternal and paternal) who are ethnically Japanese and having Japanese lifestyle, including diet, as determined by participant's verbal report.
* Good health status as determined by investigator according to past medical history, clinical examination, including 12 lead ECG, vital signs (blood pressure, pulse rate, respiratory rate and body temperature) and laboratory tests at screening and inclusion.

Exclusion Criteria:

* Pregnant or breast-feeding female volunteer.
* Having acute or chronic renal insufficiency, defined as an eGFR (estimated Glomerular Filtration Rate) <90mL/min/1.73 m2, calculated by using the Japanese coefficient-modified CKD-EPI formula.
* With known contra-indication(s) to the use or with known sensitivity to one of the products under investigation or to drugs from a similar pharmaceutical class.
* With known history of severe allergic or anaphylactic reactions to any allergen including drugs and contrast agents.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Cmax | from baseline (30 minutes before injection) to 24hours post injection
  Maximum concentrations measured, value taken directly from the observed concentration-time profiles
Tmax | from baseline (30 minutes before injection) to 24hours post injection
  Time corresponding to Cmax
AUC 0-inf | from baseline (30 minutes before injection) to 24hours post injection
  Area Under the observed concentration-time Curve from zero (time of drug administration) to infinity with extrapolation of the terminal phase. It will be obtained as follows: AUC 0-inf = AUC 0-T last + (Clast / β)
t 1/2β | from baseline (30 minutes before injection) to 24hours post injection
  Terminal elimination half-life of gadopiclenol calculated as follows:
  t 1/2β = ln 2 / β
AUC extrap% | from baseline(30 minutes before injection) to 24hours post injection
  Percentage of extrapolation of AUC from the last observation (Tlast) to infinity calculated as follows:
  Percentage of extrapolation of AUC from the last observation (Tlast) to infinity calculated as follows:
  Percentage of extrapolation of AUC from the last observation (Tlast) to infinity calculated as follows:
CLT | from baseline (30 minutes before injection) to 24hours post injection
  Total Clearance, calculated as CLT = Dose /AUC 0-inf
Vdβ | from baseline (30 min before injection) to 24h post injection
  Volume of distribution, calculated as Vdβ = Dose / (AUC 0-inf x β)
Ae | Before administration and during intervals 0-6hours, 6-24hours and 24-48hours after gadopiclenol administration
  Total amount of gadopiclenol excreted in urine
CLR | Before administration and during intervals0-6hours, 6-24hours and 24-48hours after gadopiclenol administration
  Renal clearance, calculated as CLR = Ae / AUC 0-inf

CONTACTS AND LOCATIONS:
Overall Officials: Jing Hao, Study Chair — Guerbet
Locations (1):
- Hataka clinic, Fukuoka, Japan